CLINICAL TRIAL: NCT00989833
Title: A Randomised, Double Blind, Placebo Controlled, Parallel-group Study With Use of Budesonide/Formoterol "As-needed", or Terbutaline "As-needed" or Regular Use of Budesonide + Terbutaline "As-needed", in Patients With Mild Intermittent Asthma
Brief Title: Comparing Symbicort® As-Needed or Bricanyl As-Needed or Pulmicort® Once Daily + Bricanyl As-Needed in Asthma Patients
Acronym: MIA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: D5890L00032
Record Dates: First submitted 2009-09-30; First posted 2009-10-06 (Estimated); Results first posted 2012-08-14 (Estimated); Last update posted 2012-08-14 (Estimated); Status verified 2012-07

CONDITIONS: Exercise Induced Asthma
Keywords: Exercise induced asthma; Mild intermittent asthma; Exercise induced bronchoconstriction
MeSH Terms: conditions — Asthma, Exercise-Induced | interventions — Budesonide; Terbutaline; Budesonide, Formoterol Fumarate Drug Combination

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- A (Active Comparator): budesonide 400yg + terbutaline 0.4 mg as-needed
  Interventions: Drug: budesonide; Drug: terbutaline
- B (Active Comparator): placebo + terbutaline 0.4 mg as-needed
  Interventions: Drug: terbutaline
- C (Active Comparator): placebo + budesonide/formoterol 160/4.5 yg as-needed
  Interventions: Drug: budesonide/formoterol

INTERVENTIONS:
Drug: budesonide — 400 yg x 1
  Other Names: Pulmicort Turbuhaler
  Arms: A
Drug: terbutaline — 0.4 mg as-needed
  Other Names: Bricanyl Turbuhaler
  Arms: A; B
Drug: budesonide/formoterol — 160/4.5 yg as-needed
  Other Names: Symbicort Turbuhaler
  Arms: C

SUMMARY:
1. The primary objective of this study is:

   * To evaluate the magnitude of the protective effect of the combination of budesonide and formoterol on an as-needed basis compared to the use of terbutaline as-needed on exercise induced bronchoconstriction in adults and adolescents with mild intermittent asthma
2. The secondary objectives of this study are:

   * To evaluate the magnitude of the protective effect of the combination of budesonide and formoterol as-needed compared to regular once daily use of budesonide plus terbutaline as-needed on exercise induced bronchoconstriction in adults and adolescents with mild intermittent asthma
   * To evaluate safety of budesonide/formoterol as-needed, terbutaline as-needed and regular use of budesonide + terbutaline as-needed as terms of adverse event

ELIGIBILITY:
Inclusion Criteria:

* History of exercise induced asthma
* Maximum 4 asthmatic episodes per week requiring use of reliever medication

Exclusion Criteria:

* No previous treatment with inhaled oral corticosteroids during the last month before randomisation
* Suspected poor capability to follow instructions, ie to exercise 3-4 times a week

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2009-09; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kjell Larsson, Professor, Principal Investigator — AstraZeneca MC Sweden; Georgios Stratelis, Study Director — AstraZeneca MC Sweden
Locations (10):
- Norway (2):
  - Research Site, Oslo
  - Research Site, Trondheim
- Sweden (8):
  - Research Site, Gothenburg
  - Research Site, Huddinge
  - Research Site, Linköping
  - Research Site, Luleå
  - Research Site, Lund
  - Research Site, Skene
  - Research Site, Stockholm
  - Research Site, Uppsala

REFERENCES:
- [Derived] Lazarinis N, Jorgensen L, Ekstrom T, Bjermer L, Dahlen B, Pullerits T, Hedlin G, Carlsen KH, Larsson K. Combination of budesonide/formoterol on demand improves asthma control by reducing exercise-induced bronchoconstriction. Thorax. 2014 Feb;69(2):130-6. doi: 10.1136/thoraxjnl-2013-203557. Epub 2013 Oct 3. PMID 24092567

RESULTS

PARTICIPANT FLOW:
Recruitment Details: On Visit 1, a total of 189 patients, aged 12-67, were enrolled at 10 study sites in 2 countries: Sweden and Norway. Of 189 enrolled patients, 66 patients were randomized and allocated to study treatment on Visit 3 (7 patients in Norway and 59 patients in Sweden).
Pre-assignment Details: A standardized exercise test (ECT) with duration of 6 minutes, at approximately 90% of maximal aerobic capacity (as defined on Visit 1) was performed on a treadmill while breathing dry air on Visit 2. Patients with exercised induced bronchoconstriction (defined as fall in FEV1 ≥ 10% ) could be randomized on Visit 3.
Groups:
- Budesonide/Terbutaline: Budesonide once daily and terbutaline before exercise and as needed
- Terbutaline: Placebo budesonide once daily and terbutaline before exercise and as needed
- Budesonide/Formoterol: Placebo budesonide once daily and budesonide/formoterol before exercise and as needed
Period: Overall Study
Arm/Group | Budesonide/Terbutaline | Terbutaline | Budesonide/Formoterol
Started | 21 | 22 | 23
Completed | 19 | 19 | 21
Not Completed | 2 | 3 | 2
Not completed — Lost to Follow-up | 0 | 1 | 0
Not completed — Protocol Violation | 1 | 2 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 1
Not completed — Incorrectly randomized | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Budesonide/Terbutaline | Terbutaline | Budesonide/Formoterol | Total
Number analyzed (Participants) | 21 | 22 | 23 | 66
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 2 | 5 | 5 | 12
  Between 18 and 65 years | 18 | 16 | 18 | 52
  >=65 years | 1 | 1 | 0 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 6 | 14 | 30
  Male | 11 | 16 | 9 | 36

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in Maximum Post-exercise Forced Expiratory Volume in One Second (FEV1) Fall After 6 Weeks
Description: FEV1
Time Frame: Baseline and Visit 6
Population: The Full Analysis Set (FAS) comprises all randomized patients regardless of whether they took IP or not and for whom data had been recorded in the CRF after randomization.
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Budesonide/Terbutaline | Terbutaline | Budesonide/Formoterol
Number analyzed (Participants) | 20 | 21 | 21
Percent change | -5.85 (6.50) | 0.61 (10.92) | -5.24 (9.64)

2. Secondary Outcome: Percent Change in Maximum Post-exercise FEV1 Fall After 3 Weeks
Description: FEV1
Time Frame: Baseline and 3 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Budesonide/Terbutaline | Terbutaline | Budesonide/Formoterol
Number analyzed (Participants) | 20 | 21 | 21
Percent change | -4.07 (5.56) | -1.19 (8.03) | -3.81 (8.68)

3. Secondary Outcome: Bronchial Responsiveness to Mannitol
Description: Change in cumulative Mannitol dose in mg in patients with a positive mannitol provocation test at baseline (PD15)
Time Frame: Baseline and 6 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Budesonide/Terbutaline | Terbutaline | Budesonide/Formoterol
Number analyzed (Participants) | 11 | 6 | 5
mg | 67.26 (141.98) | -6.15 (95.10) | 151.87 (141.09)

4. Secondary Outcome: Concentration of Exhaled Nitric Oxide
Time Frame: 6 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ppb
Arm/Group | Budesonide/Terbutaline | Terbutaline | Budesonide/Formoterol
Number analyzed (Participants) | 19 | 18 | 21
ppb | 25.9 (20.1) | 35.5 (36.6) | 24.4 (22.4)

5. Secondary Outcome: Use of as Needed Medication
Description: Mean number of as needed inhalations taken before exercise
Time Frame: 6 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: number of inhalations per day
Arm/Group | Budesonide/Terbutaline | Terbutaline | Budesonide/Formoterol
Number analyzed (Participants) | 20 | 20 | 21
number of inhalations per day | 0.6 (0.2) | 0.8 (0.5) | 0.7 (0.5)

6. Secondary Outcome: Asthma Control Measured by a 5-item Asthma Control Questionnaire (ACQ5)
Description: Change in overall ACQ5. ACQ5 measures asthma control and a lower values shows a better asthma control, a higher value is worse. A decrease in the ACQ5 shows an improvement during the treatment period. Range of ACQ5 is 0-5, with 0 as the best value and 5 as the worst value. Further information at www.qoltech.co.uk.
Time Frame: Baseline e and 6 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Budesonide/Terbutaline | Terbutaline | Budesonide/Formoterol
Number analyzed (Participants) | 20 | 21 | 22
units on a scale | -0.3 (0.7) | -0.2 (0.8) | -0.4 (0.7)

7. Secondary Outcome: Diary Recording of Asthma Symptoms
Description: Asthma symptoms during days with exercise
Time Frame: 6 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percent of exercise days
Arm/Group | Budesonide/Terbutaline | Terbutaline | Budesonide/Formoterol
Number analyzed (Participants) | 20 | 20 | 21
Percent of exercise days | 51.1 (30.5) | 50.9 (36.6) | 49.8 (26.1)

8. Secondary Outcome: Number of Participants With an Adverse Event During the Study
Time Frame: 6 weeks
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Budesonide/Terbutaline | Terbutaline | Budesonide/Formoterol
Number analyzed (Participants) | 21 | 22 | 23
Participants | 13 | 13 | 13

ADVERSE EVENTS:
Arm/Group | Budesonide/Terbutaline | Terbutaline | Budesonide/Formoterol
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/22 | 0/23
Other Adverse Events (participants affected / at risk) | 7/21 | 10/22 | 9/23
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Budesonide/Terbutaline (N=21) | Terbutaline (N=22) | Budesonide/Formoterol (N=23)
Common cold (Infections and infestations) | 5 | 7 | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 1
Gastroenteritis (Gastrointestinal disorders) | 1 | 0 | 3
Sore throat (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 4
Headache (General disorders) | 1 | 2 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 2
Slight Fever (General disorders) | 0 | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less